CLINICAL TRIAL: NCT06412302
Title: No-Whey: High Protein Dairy and Resistance Exercise for the Improvement of Body Composition and Muscle Function in the Elderly
Brief Title: High Protein Dairy Products and Resistance Exercise in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de O´Higgins (Other)
Collaborators: Instituto de Nutrición y Tecnología de los Alimentos (Other); Geroscience Center for Brain Health and Metabolism (Gero) (Other Government); Motion Health and Performance Center (Unknown)
Responsible Party: Principal Investigator, Matias Monsalves Álvarez, Principal Investigator, Universidad de O´Higgins
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 027-2023
Record Dates: First submitted 2024-05-06; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Dairy Products; Whey Protein; Resistance Training; Older Adults

STUDY DESIGN:
Intervention Model Description: The PY group will be provided with two yogurts and 50 of water (220g per serving, containing 24.6g protein, 1.4g fat, and 16.6 carbohydrates), while the WP will be provided with a shake with water (25g per serving containing; 25g protein, 0g fat, and 1g carbohydrates, dissolved in water), immediately after the exercise session which a trainer will monitor. Both groups will submit to a resistance training group every 8 weeks.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey Protein+Resistance Training (Experimental): Participants will undergo 8 weeks of resistance training and receive a whey protein shake after each exercise session.
  Interventions: Other: Whey Protein+Resistance Training
- Protein Yogurt+Resistance Training (Experimental): Participants will undergo 8 weeks of resistance training and receive a yogurt shake after each exercise session.
  Interventions: Other: High protein yogurt+Resistance Training

INTERVENTIONS:
Other: Whey Protein+Resistance Training — WP group received 25g protein on one scoop of Whey Protein Isolate (Iso100 Dymatize) with 8 weeks of resistance training 3 days a week.
  Other Names: WP
  Arms: Whey Protein+Resistance Training
Other: High protein yogurt+Resistance Training — PY group received 24.6g protein on two High Protein yogurts (Lonco Leche) with 8 weeks of resistance training 3 days a week.
  Other Names: PY
  Arms: Protein Yogurt+Resistance Training

SUMMARY:
Protein supplementation is one of the main recommendations for regular endurance physical exercise (RT). In older people, the need for protein increases particularly in the face of physiological and pathophysiological changes associated with the loss of muscle tissue and function, so protein intake becomes more relevant in this population. Fermented dairy products such as yogurt, and especially those with an extra protein content, have increased their popularity and consumption in the national market. Their nutritional composition is of particular interest, given their amino acid profile and in particular their high Leucine content, which could be compared with the classic protein supplements recommended for muscle gain and recovery. Objective: To analyze the effect on body composition, lipid profile, physical condition and muscle functionality induced by the intake of high protein yogurts versus Whey protein together with a muscular resistance program in elderly people. Hypothesis: The intake of high protein yogurts will lead to equal or greater gains in muscle mass, physical condition and functionality than those obtained with the intake of Whey protein together with resistance training in elderly people.Methodology: 16 healthy, lactose intolerant free, older (60-75 years old) subjects will be recruited to perform 8 weeks of muscular resistance training (RT) 3 times per week, who will be randomly supplemented with high protein yogurt (PY) or Whey protein (WP). At baseline and at the end of the intervention, body composition will be assessed by DEXA, muscle strength, maximal oxygen consumption and lipid profile. Expected Results: The YPRT group is expected to achieve similar or greater increases in muscle strength, fat-free mass, lipid profile and decrease in fat mass than the WP group.

ELIGIBILITY:
Inclusion Criteria:

* >60 years
* Less than 1 hour of exercise a week

Exclusion Criteria:

* Lactose Intolerant
* Smoking
* Type 1 or 2 Diabetes
* Alcohol intake
* Currently taking protein, high protein yogurts, creatine, HMB or any other supplement that aims to improve muscle mass

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Body Composition | From Baseline, up to 56 days
  Changes in weight, total fat mass, total skeletal muscle mass, segmental fat and muscle mass
Blood Lipids | From Baseline, up to 56 days
  Changes on Serum Triglycerides, Total Cholesterol, and High Density Cholesterol (mmol/L)
Muscle Strength | From Baseline, up to 56 days
  Determine by Isometric mid-tight pull (Newton, N)
Handgrip | From Baseline, up to 56 days
  Handgrip Strength measured on left and right hand (kg)
Time Up and Go | From Baseline, up to 56 days
  Length of time from sitting-walk-sit (seconds)
Isokinetic Muscle Strength | From Baseline, up to 56 days
  Maximal peak torque from left and right quadriceps and hamstrings (N/m)
Aerobic Capacity | From Baseline, up to 56 days
  Maximal Oxygen Consumption determine by the volume of oxygen (L/min)obtained on a incremental test
Resting Metabolic Rate | From Baseline, up to 56 days
  Determine by indirect calorimetry (kcal/d)
Evaluation of the intestinal microbiota | From Baseline, up to 56 days
  Fecal microbiota analysis based on the 16S ribosomal RNA (rRNA) sequencing pre- and post-dietary intervention.

SECONDARY OUTCOMES:
Food Consumption | From Baseline, up to 56 days
  24h food recall
Evaluation of liver characteristics profile | From Baseline, up to 56 days
  Uric acid, BUN, Albumin, Creatinine aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), gamma-glutamyltransferase (GGT) after every intervention and wash-out in plasma (mmol/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Motion Health and Performance Center, Santiago, Chile